CLINICAL TRIAL: NCT02459548
Title: Validation of a Programme of Treatment and Follow-Up for Obstructive Sleep Apnea (OSA) Patients to be Applied by General Practitioners (GPs). Collaborative Network System Between GPs, CPAP Provider Enterprise and Sleep Specialists
Brief Title: Continuous Positive Airway Pressure (CPAP) for Primary Care
Acronym: CPAP-SU-MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Spain:Health Department. Basque Government. (Unknown); Linde Health Care (Other)
Responsible Party: Principal Investigator, Joaquin Duran-Cantolla, MD, Joaquin Duran-Cantolla, MD Hospital Universitario Araba, Vitoria-Gasteiz (Spain), Hospital Universitario Araba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2010111082
Record Dates: First submitted 2015-04-01; First posted 2015-06-02 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: OSA
Keywords: OSA; CPAP treatment; Primary care; Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care Group (Experimental): This group will be follow up in Primary Care at 1, 3 and 6 month. At each visit patients receive advice on CPAP treatment, management of adverse effects associated with CPAP, making anthropometric and blood pressure measurements and also were asked to complete questionnaires.
  Interventions: Other: Follow up in Primary Care Group
- Sleep Unit Group (Other): This group will be follow up in Sleep unit at 1, 3 and 6 month. At each visit patients receive advice on CPAP treatment, management of adverse effects associated with CPAP, making anthropometric and blood pressure measurements and also were asked to complete questionnaires.
  Interventions: Other: Follow up in Sleep Unit Group

INTERVENTIONS:
Other: Follow up in Sleep Unit Group — Compare the results of a program of treatment and follow-up by Primary Care in patients with obstructive sleep apnea on CPAP treatment, versus the usual practice of control by the Sleep Unit.
  Arms: Sleep Unit Group
Other: Follow up in Primary Care Group — Compare the results of a program of treatment and follow-up by Primary Care in patients with obstructive sleep apnea on CPAP treatment, versus the usual practice of control by the Sleep Unit.
  Arms: Primary Care Group

SUMMARY:
The objective of the study is to compare the results of a follow-up and treatment coordinate and interactive program performed by the General Practitioners (GP) for Obstructive Sleep Apnea (OSA) patients treated with positive continuous pressure (CPAP) vs. usual control by sleep specialists from the sleep unit.

METHODOLOGY: DESIGN: Randomized comparative study. It will include patients with diagnosis of severe OSA that should start treatment with CPAP. Participating center is Hospital Universitario Araba in Vitoria-Gasteiz (Spain). These patients will be randomized to two monitoring groups : 1 monitoring in the sleep unit; 2: monitoring in primary care consultations by the General Practitioners (GP), once the OSA diagnosis has been made and it was indicated the treatment with CPAP.

Patients will be carried out in both groups the same follow-up visits in two study arms: basal, 1 month, 3 month and 6 months. PRIMARY OUTCOME: To compare the objective CPAP compliance treatment in the two study groups, so that use >= 4h/day is defined as good adherence to the treatment. SECONDARY OUTCOMES: 1)To evaluate the level of patient's satisfaction by visual-analogical scales and quality of life tests; 2) to establish the clinical improvement by somnolence and sleep scales; 3) To determine the numbers of CPAP complications, type, severity and duration; 4) To figure-out the level of take care of the CPAP machine, substitutions and complements, assistance and technical incidents; 5) Cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Patients with OSA diagnosis performed in the sleep unit
* Written informed consent signed.

Exclusion Criteria:

* Previous CPAP treatment for OSA diagnosis
* Psycho-physical inability to complete questionnaires
* Presence of any previously diagnosed sleep disorders: narcolepsy, insomnia, chronic sleep deprivations, regular use of hypnotic or sedative medications nad restless leg syndrome
* Patients with respiratory diseases (overlap syndrome, hypoventilation, restrictive diseases)
* A medical history that may interfere with the study objectives or, in the opinion of the investigator, compromise the conclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of hours of use per day of CPAP | Six month
  Compare the objective CPAP compliance treatment in the two study groups.

SECONDARY OUTCOMES:
Level of clinical improvement evaluated through the Epworth Sleep Scale | At baseline and at 6 month of follow-up
  Evaluate the level of clinical improvement from the start of treatment until 6 months by the changes in the Epworth Sleep Scale
Patient satisfaction (visual-analogical scale) | Six month
  Evaluate the level of patient's satisfaction by visual-analogical scale.
Adverse events (number of CPAP complications) | Six month
  Determine the number of CPAP complications (secondary effects).
Quality of life (EuroQOL test) | Baseline and at 6 month of follow up
  Evaluate by EuroQOL test
Comorbidity index (Charlson index) | Six month
  Charlson index
Blood pressure | Six month
  Blood pressure measurements
Cost-effectiveness analysis | Six month
  Cost-efficacy evaluation

OTHER OUTCOMES:
Anthropometric variables (Body mass index) | Six month
  Body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Duran-Cantolla, MD, Principal Investigator — Hospital Universitario Araba
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Araba, Spain